CLINICAL TRIAL: NCT01239875
Title: LS1081, "A Pilot Study of Dendritic Cell Therapy Delivered Intratumorally After Cryoablation or Intradermally for Patients With B-Cell Non-Hodgkin's Lymphoma"
Brief Title: Vaccine Therapy With or Without Cryosurgery in Treating Patients With Residual, Relapsed, or Refractory B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LS1081; NCI-2010-02003 (Registry Identifier: NCI-CTRP); LS1081 (Other: Mayo Clinic Cancer Center & SPORE); 10-003023 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2010-10-27; First posted 2010-11-11 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2019-01

CONDITIONS: Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Adult Diffuse Mixed Cell Lymphoma; Adult Diffuse Small Cleaved Cell Lymphoma; Adult Grade III Lymphomatoid Granulomatosis; Adult Immunoblastic Large Cell Lymphoma; Adult Lymphoblastic Lymphoma; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3 Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia With Nodal Disease
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cryotherapy; Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Patients receive pneumococcal polyvalent vaccine intramuscularly in weeks -4, 2, and 10. Patients undergo cryoablation followed by dendritic cell vaccine (CA-DC) intratumorally in weeks 0, 2, 4, 6, 10, 14, 18, and 22.
  Interventions: Biological: dendritic cell vaccine therapy; Procedure: cryotherapy; Biological: pneumococcal polyvalent vaccine; Other: laboratory biomarker analysis; Other: immunoenzyme technique; Other: immunohistochemistry staining method
- Arm B (Experimental): Patients receive pneumococcal polyvalent vaccine as in arm A. Patients also receive autologous dendritic cell-tumor fusion vaccine (TL-DC) intradermally in weeks 0, 2, 4, 6, 10, 14, 18, and 22.
  Interventions: Biological: dendritic cell vaccine therapy; Biological: pneumococcal polyvalent vaccine; Other: laboratory biomarker analysis; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Biological: autologous dendritic cell-tumor fusion vaccine

INTERVENTIONS:
Biological: dendritic cell vaccine therapy — Given intratumorally
Procedure: cryotherapy — Undergo cryoablation
  Arms: Arm A
Biological: pneumococcal polyvalent vaccine — Given intramuscularly
  Other Names: Pneumovax 23; Pnu-Imune 23
Other: laboratory biomarker analysis — Correlative studies
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Biological: autologous dendritic cell-tumor fusion vaccine — Given intradermally
  Arms: Arm B

SUMMARY:
RATIONALE: Vaccines, such as dendritic cell therapy (DC) made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells. Cryosurgery kills cancer cells by freezing them. Giving vaccine therapy together with cryosurgery may kill more tumor cells. PURPOSE: This clinical trial studies giving vaccine therapy together with or without cryosurgery in treating patients with B-cell Non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Evaluation of safety and tolerability as measured by the incidence of significant toxicity of an autologous DC vaccine injection into a cryoablated tumor site (Arm A). II. Evaluation of safety and tolerability as measured by the incidence of significant toxicity of an autologous mature DC vaccine + tumor lysate generated in vitro and delivered intradermally (ID) (Arm B). SECONDARY OBJECTIVES: I. For cryoablation candidates: To assess feasibility, overall response rate, clinical benefit rate, time to response, and duration of response (Arm A). II. For patients receiving ID vaccine without cryoablation: To assess feasibility, clinical response rate, time to response, and duration of response (Arm B). TERTIARY OBJECTIVES: I. For cryoablation candidates: To assess the change over time in non-cryoablated nodes selected as the index lesions (Arm A). II. For patients receiving ID vaccine without cryoablation: To assess the change over time in measurable nodes selected as the index lesions (Arm B). III. To monitor patients' immune response after vaccine therapy. IV. Assess the immune response to Prevnar in cancer patients. V. Assess the effect of DC vaccination on presence of myeloid suppressors. VI. Assess the effect of tumor antigen delivery methods (in vivo DC into cryoablated tumor vs. ID injection of in vitro generated DC + lysate) on T cell response. OUTLINE: Patients are assigned to 1 of 2 treatment arms. In both arms, treatment continues in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 3 months for 1 year, and then every 6 months for up to 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of biopsy-proven B-cell non-Hodgkin's lymphoma, excluding chronic lymphocytic leukemia, primary CNS lymphoma and Burkitt's lymphoma.
* Patient must have at least 2 measurable lesions that are >= 1.5cm in one dimension. One of the lesions, must meet additional criteria a or b depending on the treatment arm. a) For Arm A, patient must have at least one lesion that is >= 2.0cm and is amenable to image-guided cryoablation and multiple vaccine injections as determined by Interventional Radiology (including tumors that can be safely accessed using imaging guidance and treated with minimal risk to adjacent structures). b) For Arm B, patient must have one lesion that can be excised for in vitro vaccine preparation.
* ECOG Performance Status (PS) 0, 1, 2
* Absolute neutrophil count > 1000/uL
* Absolute lymphocyte count > 500/uL
* PLT >= 100,000/uL
* HgB >= 8.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN, the direct bilirubin must be normal
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willingness to return to a Lymphoma SPORE enrolling institution for follow-up
* Patient willing to provide tissue and blood samples for research purposes

Exclusion Criteria:

* Pregnant women
* Nursing women
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Patients known to be HIV positive
* Serious non-malignant disease such as active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations or other conditions which in the opinion of the investigator would compromise protocol objectives
* Receiving any other investigational agent considered as a treatment for the primary neoplasm
* History of other primary malignancy requiring systemic treatment within 6 months of protocol enrollment
* Patients must not have another active malignancy requiring treatment
* Patients must not be receiving chemotherapy or immunotherapy for another cancer
* Prior allogeneic bone marrow or peripheral blood stem cell transplantation
* Prior autologous bone marrow or peripheral blood stem cell support within 1 year
* Major surgery other than diagnostic surgery =< 4 weeks
* History of hypersensitivity and anaphylactoid reactions to pneumococcal vaccine or any component of the formulation, including diphtheria toxoid
* Active autoimmune disease such as Crohn's disease, rheumatoid arthritis, Sjogrens' disease, systemic lupus erythematosis, or similar conditions
* Coagulopathy, including the use of Coumadin or heparin anticoagulants that cannot be discontinued for the cryoablation procedure (NOTE: Heparin for line patency without detectable lab abnormalities for coagulation will be allowed)
* Patients must be off corticosteroids for at least 2 weeks prior to registration (this includes oral, IV, subcutaneous, or inhaled route of administration); patients on chronic corticosteroid for adrenal insufficiency or other reasons may enroll if they receive less than 10 mg/day of prednisone (or equivalent)
* Patients with active CNS malignancy are not eligible for this trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2015-11-24 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Incidence of significant toxicity as assessed by the CTEP Active Version CTCAE | At day 1 of each course beginning in week 2, every 3 months for 1 year, and during documented progressive disease

SECONDARY OUTCOMES:
Overall response rate | At week 4 (arm A) or 2 (arm B) and then every 3 months for 1 year starting at week 10
Feasibility as estimated by the number of patients receiving at least one dose of tumor antigen loading and vaccine delivery divided by the number receiving leukapheresis | Up to 2.5 years
Clinical benefit rate as estimated by the number of patients with an objective status of stable disease (SD) or an objective status of CR or PR | For at least 12 months
Time to response | From the date of initiation of vaccination treatment to the date at which the patient's objective status is first noted to be either a CR or PR
Duration of response | From the date at which the patient's objective status is first noted to be either a CR or PR to the earliest date progression is documented
Percent change from baseline in index lesion measurements as a marker of distant immune and treatment response | At day 1 of courses 1-4 (arm A) and 1-6 (arm B)
Change in immunologic correlates before and after vaccination treatment | At day 1 of each course beginning in week 2, every 3 months for 1 year, and during documented progressive disease
Correlation of immunologic markers with cancer and treatment-related outcomes (e.g., response, toxicities) | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lin, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States